CLINICAL TRIAL: NCT01289782
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety and Tolerability of TMC435 vs Placebo as Part of a Treatment Regimen Including Peginterferon α-2a and Ribavirin in Treatment-naïve, Genotype 1 Hepatitis Cinfected Subjects
Brief Title: An Efficacy, Safety, and Tolerability Study of TMC435 in Treatment-naive, Genotype 1 Hepatitis C-infected Patients
Acronym: QUEST-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017386; TMC435-TiDP16-C208 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2011-01-07; First posted 2011-02-04 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435; HCV; Hep C; Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMC435 (Experimental): TMC435 150 mg capsule once daily for 12 weeks in addition to peginterferon alpha-2a (PegIFN alpha-2a) and ribavirin (RBV) for 24 or 48 weeks
  Interventions: Drug: TMC435; Drug: Peginterferon alpha-2a (PegIFN alpha-2a); Drug: Ribavirin (RBV)
- Placebo (Placebo Comparator): Placebo 150 mg capsule once daily for 12 weeks in addition to PegIFNα-2a and RBV for 48 weeks
  Interventions: Drug: Placebo; Drug: Peginterferon alpha-2a (PegIFN alpha-2a); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Placebo — 150 mg capsule once daily for 12 weeks in addition to PegIFN alpha-2a and RBV for 48 weeks
  Arms: Placebo
Drug: TMC435 — 150 mg capsule once daily for 12 weeks in addition to PegIFN alpha-2a and RBV for 24 or 48 weeks
  Arms: TMC435
Drug: Peginterferon alpha-2a (PegIFN alpha-2a) — One subcutaneous (under the skin) injection containing 0.5 mL solution with 180 mcg PegIFN alpha-2a once weekly for up to 48 weeks.
  Other Names: Pegasys
Drug: Ribavirin (RBV) — 200-mg tablets of RBV (body-weight adjusted dose) taken orally (by mouth) twice daily for up to 48 weeks.
  Other Names: Copegus

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of TMC435 compared with placebo in participants who are infected with genotype 1 hepatitis C virus who have never received treatment before. Participants will also receive peginterferon alpha-2a and ribavirin as part of their treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither physician nor participants know the name of the assigned drug), placebo-controlled study of TMC435 in participants who are infected with genotype 1 hepatitis C virus (HCV), who have never received treatment for HCV infection before. Participants in this study will also receive two other drugs for their HCV infection called peginterferon alpha-2a (PegIFN alpha-2a) and ribavirin (RBV). The purpose of the study is to investigate if TMC435 is superior to placebo in reducing plasma levels of HCV ribonucleic acid (RNA) to an undetectable level 12 weeks after the end of treatment. For the first 12 weeks, participants will take either TMC435 or placebo, plus PegIFNα-2a and RBV. For the next 12 weeks, participants will take PegIFN alpha-2a and RBV only. After that, some participants will continue to take PegIFN alpha-2a and RBV for up to 24 additional weeks and some will stop taking PegIFN alpha-2a and RBV depending on response-guided treatment criteria. The study doctor will inform each participant about how to take their study medication and when they should stop taking it. After a participant stops taking study medication, they will continue to come to the doctor's office for study visits until a total of 72 weeks after they enroll in the study. The total duration of the study is 78 weeks (including screening). Participants will be monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 hepatitis C infection (confirmed at screening)
* Patient has not received any prior treatment for hepatitis C
* Patient must have had a liver biopsy within 3 years before screening (or between the screening and baseline visit) showing chronic hepatitis C infection
* Must agree to use 2 forms of effective contraception throughout study (both males and females)

Exclusion Criteria:

* Infection with HIV or non genotype 1 hepatitis C
* Liver disease not related to hepatitic C infection
* Hepatic decompensation
* Significant laboratory abnormalities or other active diseases
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (62):
- United States (22):
  - Dothan, Alabama
  - Hoover, Alabama
  - Phoenix, Arizona
  - Bakersfield, California
  - Coronado, California
  - Long Beach, California
  - San Diego, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Miami, Florida
  - Chicago, Illinois
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
- Australia (6):
  - Darlinghurst
  - Fitzroy
  - Kingswood
  - Melbourne
  - Sydney
  - Wolloongabba
- Canada (4):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (4):
  - Berlin
  - Heidelberg
  - Kiel
  - Tübingen
- Mexico (3):
  - Guadalajara
  - Mex Ctity
  - Monterrey
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton
- San Juan, Puerto Rico
- Bucharest, Romania
- Russia (5):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Samara
  - Smolensk
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Ukraine (4):
  - Donetsk
  - Kiev
  - Kyiv
  - Vinnytsia
- United Kingdom (5):
  - Derby
  - Liverpool
  - London
  - Nottingham
  - Plymouth

REFERENCES:
- [Derived] Lenz O, Verbinnen T, Fevery B, Tambuyzer L, Vijgen L, Peeters M, Buelens A, Ceulemans H, Beumont M, Picchio G, De Meyer S. Virology analyses of HCV isolates from genotype 1-infected patients treated with simeprevir plus peginterferon/ribavirin in Phase IIb/III studies. J Hepatol. 2015 May;62(5):1008-14. doi: 10.1016/j.jhep.2014.11.032. Epub 2014 Nov 28. PMID 25445400
- [Derived] Jacobson IM, Dore GJ, Foster GR, Fried MW, Radu M, Rafalsky VV, Moroz L, Craxi A, Peeters M, Lenz O, Ouwerkerk-Mahadevan S, De La Rosa G, Kalmeijer R, Scott J, Sinha R, Beumont-Mauviel M. Simeprevir with pegylated interferon alfa 2a plus ribavirin in treatment-naive patients with chronic hepatitis C virus genotype 1 infection (QUEST-1): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2014 Aug 2;384(9941):403-13. doi: 10.1016/S0140-6736(14)60494-3. Epub 2014 Jun 4. PMID 24907225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 18 January 2011 to 29 January 2013. The study was conducted at 71 sites in 13 countries.
Pre-assignment Details: 395 participants were randomly allocated to the 2 treatment arms. 394 participants received at least 1 dose of study medication and were included in the intent-to-treat analysis set.
Groups:
- TMC435 150mg 12Wks PR24/48: Participants were given TMC435 150 mg once daily plus peginterferon alpha-2a (PegIFN alpha-2a) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFN alpha-2a (P) and RBV (R) until Week 24 (PR24). Treatment was to be stopped at Week 24 for participants who achieved HCV RNA < 25 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA at Week 12. Other participants continued PR until Week 48 (PR48).
- PBO 12Wks PR48: Participants were given placebo (PBO) once daily plus peginterferon alpha-2a (PegIFN alpha-2a) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFN alpha-2a (P) and RBV (R) until Week 48 (PR 48).
Period: Overall Study
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Started | 264 | 130 (Not including 1 participant was randomized to this group, but never received treatment.)
Completed | 239 | 118
Not Completed | 25 | 12
Not completed — Lost to Follow-up | 14 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Sponsor's Decision | 1 | 0
Not completed — Reason not specified | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48 | Total
Number analyzed (Participants) | 264 | 130 | 394
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 68] | 48 [20 to 66] | 48 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 56 | 172
  Male | 148 | 74 | 222

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Planned End of Treatment (SVR12)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR12, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid 12 weeks after planned end of treatment.
Time Frame: Week 36 or Week 60
Population: The intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) was used for all analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 79.5 | 50
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Null hypothesis: There is no difference in proportions of SVR12 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR12 = 29.3, 95% CI 2-sided [20.1 to 38.6]

2. Secondary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response at Week 72 (SVRW72)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVRW72, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels at end of treatment (EOT) and at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 78.4 | 49.2
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; There is no difference in proportions of SVRW72 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVRW72 = 28.9, 95% CI 2-sided [19.6 to 38.2]

3. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 24 Weeks After the Planned End of Treatment (SVR24)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR24, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels 24 weeks after planned end of treatment.
Time Frame: Week 48 or Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 79.5 | 49.2
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; There is no difference in proportions of SVR24 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR24 = 30.1, 95% CI 2-sided [20.8 to 39.3]

4. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 4 Weeks After the Planned End of Treatment (SVR4)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR4, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels 4 weeks after planned end of treatment.
Time Frame: Week 28 or Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 82.2 | 56.2
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; There is no difference in proportions of SVR4 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR4 = 25.8, 95% CI 2-sided [16.8 to 34.8]

5. Secondary Outcome: Change From Baseline in log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The table below shows the change from baseline in log10 HCV RNA levels.
Time Frame: Day 3, Week 1, Week 4, Week 12, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
log10 IU/mL
  Day 3 | -3.52 (0.0459) | -0.93 (0.0774)
  Week 1 | -4.47 (0.0512) | -1.08 (0.0835)
  Week 4 | -5.22 (0.0552) | -2.56 (0.1434)
  Week 12 | -5.34 (0.0524) | -4.18 (0.1510)
  Week 24 | -5.32 (0.0604) | -4.89 (0.1289)
  Week 48 | -5.33 (0.2605) | -5.23 (0.1670)

6. Secondary Outcome: Actual Values of log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The table below shows actual values of log10 HCV RNA levels.
Time Frame: Day 3, Week 1, Week 4, Week 12, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
log10 IU/mL
  Day 3 | 2.914 (0.052) | 5.351 (0.104)
  Week 1 | 1.973 (0.052) | 5.202 (0.114)
  Week 4 | 1.223 (0.049) | 3.723 (0.159)
  Week 12 | 1.090 (0.041) | 2.111 (0.155)
  Week 24 | 1.113 (0.050) | 1.334 (0.110)
  Week 48 | 0.993 (0.039) | 0.961 (0.006)

7. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response at All Time Points
Description: The table below shows the percentage of participants with Hepatitis C virus (HCV) ribonucleic acid (RNA) plasma levels below the limit of detection (ie, <25 IU/mL undetectable), the percentage of participants with a HCV RNA plasma level below the limit of quantification (ie, < 25 IU/mL detectable or undetectable), the percentage of participants with plasma levels of HCV RNA <100 IU/mL, the percentage of participants with virologic responses of a greater than or equal to 2 log10 change from baseline in plasma levels of HCV RNA.
Time Frame: Day 3, Week 1, Week 2, Week 8, Week 16, Week 20, Week 28, Week 36, and Week 42
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants
  Day 3:<25 IU/mL undetectable | 0.4 | 0.8
  Week 1:<25 IU/mL undetectable | 6.6 | 0.8
  Week 2:<25 IU/mL undetectable | 35.8 | 2.3
  Week 8:<25 IU/mL undetectable | 90.0 | 26.2
  Week 16:<25 IU/mL undetectable | 93.8 | 69.2
  Week 20:<25 IU/mL undetectable | 93.4 | 78.2
  Week 28:<25 IU/mL undetectable | 90.9 | 96.3
  Week 36:<25 IU/mL undetectable | 90.9 | 100.0
  Week 42:<25 IU/mL undetectable | 90.9 | 98.7
  Day 3:<25 IU/mL undetectable/detectable | 2.4 | 0.8
  Week 1:<25 IU/mL undetectable/detectable | 36.8 | 2.3
  Week 2:<25 IU/mL undetectable/detectable | 76.7 | 6.3
  Week 8:<25 IU/mL undetectable/detectable | 94.0 | 40.5
  Week 16:<25 IU/mL undetectable/detectable | 95.4 | 82.7
  Week 20:<25 IU/mL undetectable/detectable | 95.0 | 84.2
  Week 28:<25 IU/mL undetectable/detectable | 100.0 | 98.8
  Week 36:<25 IU/mL undetectable/detectable | 100.0 | 100.0
  Week 42:<25 IU/mL undetectable/detectable | 100.0 | 100.0
  Day 3:<100 IU/mL | 11.4 | 1.6
  Week 1:<100 IU/mL | 62.8 | 3.1
  Week 2:<100 IU/mL | 85.2 | 7.8
  Week 8:<100 IU/mL | 94.8 | 46.0
  Week 16:<100 IU/mL | 96.7 | 84.6
  Week 20:<100 IU/mL | 96.7 | 86.1
  Week 28:<100 IU/mL | 100.0 | 98.8
  Week 36:<100 IU/mL | 100.0 | 100.0
  Week 42:<100 IU/mL | 100.0 | 100.0
  Day 3:> or = 2 log10 change from baseline | 95.3 | 13.3
  Week 1:> or = 2 log10 change from baseline | 98.1 | 20.2
  Week 2:> or = 2 log10 change from baseline | 98.8 | 35.2
  Week 8:> or = 2 log10 change from baseline | 98.4 | 80.2
  Week 16:> or = 2 log10 change from baseline | 100.0 | 99.0
  Week 20:> or = 2 log10 change from baseline | 98.3 | 97.0
  Week 28:> or = 2 log10 change from baseline | 100.0 | 97.5
  Week 36:> or = 2 log10 change from baseline | 100.0 | 98.7
  Week 42:> or = 2 log10 change from baseline | 100.0 | 98.7

8. Secondary Outcome: The Percentage of Participants Achieving a Rapid Virologic Response (RVR)
Description: The table below shows the percentage of participants in each treatment group who achieved a RVR, defined as having undetectable plasma Hepatitis C virus ribonucleic acid levels after receiving 4 weeks of treatment.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 79.5 | 11.8

9. Secondary Outcome: The Percentage of Participants Achieving a Early Virologic Response (EVR)
Description: The table below shows the percentage of participants who achieved an EVR, defined as having a change from baseline in plasma Hepatitis C virus ribonucleic acid of greater than or equal to 2 log10 at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 99.2 | 85.2

10. Secondary Outcome: The Percentage of Participants Achieving a Complete Early Virologic Response (cEVR)
Description: The table below shows the percentage of participants in each treatment group who had a cEVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 92.8 | 50.8

11. Secondary Outcome: The Percentage of Participants Achieving a Extended Rapid Virologic Response (eRVR)
Description: The table below shows the percentage of participants in each treatment group who had a eRVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 4 and 12.
Time Frame: Week 4 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 78.9 | 11.7

12. Secondary Outcome: The Percentage of Participants With <1 log10 Decrease in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) From Baseline at Week 4
Description: The table below shows the percentage of participants in each treatment group with <1 log10 HCV RNA decrease at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 0 | 15.7

13. Secondary Outcome: Percentage of Participants With in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels >1000 IU/mL at Week 4
Description: The table below shows the percentage of participants in each treatment group with HCV RNA levels >1000 IU/mL at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 4.5 | 63.8

14. Secondary Outcome: Percentage of Participants With Null Response
Description: The table below shows the percentage of participants with null response, defined as <2 log10 reduction in Hepatitis C virus ribonucleic acid at Week 12 compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 0.8 | 14.8

15. Secondary Outcome: Percentage of Participants With Partial Response
Description: The table below shows the percentage of participants with partial response, defined as greater than or equal to 2 log10 reduction in Hepatitis C virus ribonucleic acid at Week 12 compared to baseline, but not achieving undetectable HCV RNA while on treatment.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 3.2 | 13.1

16. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: The table below shows the percentage of participants with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (<25 IU/mL undetectable).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 4.9 | 7.7

17. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: The table below shows the percentage of participants with viral relapse, defined as having confirmed detectable plasma level of Hepatitis C virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (less than 25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 9.0 | 22.6

18. Secondary Outcome: Percentage of Participants Who Completed All Study Treatment at Week 24 Because of the Treatment Duration Rule
Description: The table below shows the percentage of participants in the TMC435 treatment group who met the treatment duration rule (ie, having hepatitis C virus [HCV] ribonucleic acid [RNA] levels <25 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA levels at Week 12) and completed treatment with PegIFNα-2a and RBV for 24 weeks. Participants in the TMC435 treatment group not meeting RGT criteria and participants in the placebo group were treated with PegIFNα-2a and RBV treatment for 48 weeks.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 83 | NA — RGT criteria did not apply to PBO arm

19. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: The table below shows percentage of participants with on-treatment failure defined as confirmed detectable Hepatitis C virus ribonucleic acid levels at actual end of treatment.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants | 9.1 | 33.8

20. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable or Detectable
Description: The table below shows median time in days to reach HCV RNA levels <25 IU/mL undetectable or detectable.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Days | 14 (1.25) [14 to 15] | 85 (4.89) [84 to 110]

21. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable
Description: The table below shows median time in days to reach HCV RNA levels <25 IU/mL undetectable.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Days | 28 [NA to NA] — Majority of the participants had HCV RNA undetectable for the first time at Day 28. So they all are concentrated in that time point and there is no a range around Day 28 to be drawn. | 111 [85 to 139]

22. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <100 IU/mL
Description: The table below shows median time in days to reach HCV RNA levels <100 IU/mL.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Days | 28 [NA to NA] — Majority of the participants had HCV RNA undetectable for the first time at Day 28. So they all are concentrated in that time point and there is no a range around Day 28 to be drawn. | 84 [57 to 85]

23. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <1000 IU/mL
Description: The table below shows median time in days to reach HCV RNA levels <1000 IU/mL.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Days | 4 [3 to 4] | 56.5 [56 to 57]

24. Secondary Outcome: The Percentage of Participants With Viral Breakthrough at Different Time Points
Description: The table below shows the percentage of participants at different time points with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma HCV ribonucleic acid (RNA) level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (<25 IU/mL undetectable).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Percentage of participants
  < 12 Weeks | 2.7 | 1.5
  Week 12 - Week 24 | 2.5 | 6.8
  > Week 24 | 0 | 1.2

25. Secondary Outcome: Time From End-of-treatment to Viral Relapse
Description: The table below shows the mean number of days to viral relapse, defined as participants having confirmed detectable plasma level of Hepatitis C Virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (<25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 264 | 130
Days | 100.96 (1.21) | 146.04 (5.22)

26. Secondary Outcome: The Percentage of Participants With Normalization of Alanine Aminotransferase (ALT)
Description: The percentage of participants analyzed were those with baseline ALT values out of the normal range (ie, 158 of 264 participants in the TMC435 treatment group and 89 of 130 participants in the Placebo group had ALT values at baseline that were out of the normal range.). Normalization of ALT values means that ALT values out of the normal range returned to within the normal range.
Time Frame: Up to Week 48
Population: Participants with baseline ALT values out of normal range were used for this analysis from intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication).
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 158 | 89
Percentage of participants | 81.0 | 77.5

27. Secondary Outcome: Median Time to Normalization of Alanine Aminotransferase (ALT) Levels
Description: The table below shows the median time in weeks to normalization of ALT levels.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 158 | 89
Weeks | 2.14 [1.86 to 4.00] | 8.14 [4.14 to 16.29]

28. Secondary Outcome: Plasma Concentration of TMC435: Area Under the Plasma Concentration-time Curve From the Time of Administration to 24 Hours After Dosing (AUC24h)
Description: The table below shows mean (standard deviation) values of the area under the plasma concentration-time curve from time of administration to 24 hours after dosing for TMC435 for all participants. To calculate the mean AUC 24 for the study, AUC 24 hr values were derived for each participant at each visit and then a median AUC value calcuated across all visits for each participant. The median AUC value across all visits for each participant was used to calculate the mean AUC 24 hr all participants in the study.
Time Frame: Fom the time of administration up to 24 hours after dosing at Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 259
ng*h/mL | 54795 (55627.3) [1.86 to 4.00]

29. Secondary Outcome: Plasma Concentration of TMC435: Predose Plasma Concentration (C0h)
Description: The table below shows the mean (standard deviation) values for the C0h of TMC435.To calculate the mean C0h for the study, C0h values were derived for each participant at each visit and then a median C0H value calculated across visits for each participant. The median COh value for each participant across all visits was used to calculate the mean C0h for the study.
Time Frame: Before administration of TMC435 at Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 259
ng/mL | 1825 (2306.1) [1.86 to 4.00]

30. Secondary Outcome: Plasma Concentration of TMC435: Systemic Clearance (CL)
Description: The table below shows the mean (standard deviation) values for the CL of TMC435.To calculate the mean CL for all participants in the study, CL values were first derived for each participant at each visit and then a median CL value calculated across visits for each participant. The median CL value for each participant was used to calculate the mean CL for all participants in the study.
Time Frame: Across Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 259
L/h | 5.05 (3.319) [1.86 to 4.00]

31. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for the Fatigue Severity Scale (FSS) Total Scores
Description: Study participants completed FSS questionnaires during study visits before treatment began and throughout treatment and follow-up to rate the severity and impact of fatigue they experienced in the preceding 2 weeks on their daily lives. FSS total scores are the average of nine questions with a range from 1 [no fatigue] to 7 [worst possible fatigue]. An area under the curve (AUC) analysis compared the overall severity of fatigue in each treatment group from baseline to Week 72. The null hypothesis was that there would be no difference between the treatment arms in the amount of fatigue participants experienced throughout the study resulting in equal AUC from baseline to Week 72 (AUC72) for FSS total scores. The Table below shows the lease squares (LS) mean estimates of AUC at Week 72 (as well as at Week 60) and the statistical comparison between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 130
scores on a scale*weeks
  Week 60 | 214.907 [205.9021 to 223.9115] | 235.586 [224.2016 to 246.9700]
  Week 72 | 250.522 [239.8398 to 261.2051] | 274.322 [260.8164 to 287.8279]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Fatigue Severity Score AUC60; Test type: Superiority or Other; p < 0.001, Piecewise-Linear Model Approach; Mean differences = -20.679, 95% CI 2-sided [-32.6399 to -8.7181], Standard Error of Mean 6.0979
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Fatigue Severity Score AUC72; Test type: Superiority or Other; p < 0.001, Piecewise Linear Model; Mean differences = -23.800, 95% CI 2-sided [-37.9931 to -9.6064], Standard Error of Mean 7.2358

32. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for Impairment in Overall Work Productivity Scores Due to Hepatitis C Virus (HCV) Infection and Its Treatment
Description: Impairment in overall work productivity was measured using the Work Productivity and Activity Impairment (WPAI): Hepatitis C questionnaire completed by participants during study visits throughout the study. WPAI Overall Productivity Scores ranged from 0% to 100% (higher WPAI scores indicated greater impairment in productivity). An area under the curve (AUC) analysis compared the overall WPAI Overall Work Productivity Scores in each treatment group from Baseline to Week 72. The null hypothesis was that there would be no difference between the treatment arms in the WPAI Overall Work Productivity Scores from Baseline to Week 72. The Table below shows the lease squares (LS) mean estimates of AUC at Week 72 (as well as at Week 60) in WPAI Work Productivity Scores and the statistical comparison between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 130
scores on a scale*weeks
  Week 60 | 1555.204 [1419.4052 to 1691.0026] | 1785.668 [1603.4340 to 1967.9027]
  Week 72 | 1718.241 [1558.7326 to 1877.7493] | 1966.449 [1752.2268 to 2180.6720]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Work Productivity AUC60; Test type: Superiority or Other; p = 0.030, Piecewise Linear Model; Mean differences = -230.464, 95% CI 2-sided [-438.2662 to -22.6626], Standard Error of Mean 105.9203
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Work Productivity AUC72; Test type: Superiority or Other; p = 0.047, Piecewise Linear Model; Mean differences = -248.208, 95% CI 2-sided [-492.8253 to -3.5916], Standard Error of Mean 124.6753

33. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for Impairment in Daily Activity Scores Due to Hepatitis C Virus (HCV) Infection and Its Treatment
Description: Impairment in daily activity was measured using the Work Productivity and Activity Impairment (WPAI): Hepatitis C questionnaire, Question 6. Scores ranged from 0 (no effect on activities) to 10 (completely prevented me from doing my daily activities). An area under the curve (AUC) analysis compared the impairment in daily activity scores in each treatment group from Baseline to Week 72. The null hypothesis was that there would be no difference between the treatment arms in impairment in daily activity scores from Baseline to Week 72. The Table below shows the lease squares (LS) mean estimates of AUC at Week 72 (as well as at Week 60) in the impairment in daily activity scores and the statistical comparison between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 130
scores on a scale*weeks
  Week 60 | 1514.400 [1379.7183 to 1649.0812] | 1792.460 [1611.2749 to 1973.6441]
  Week 72 | 1667.735 [1509.6180 to 1825.8526] | 1975.457 [1762.6198 to 2188.2942]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Daily Activities AUC60; Test type: Superiority or Other; p = 0.009, Piecewise linear model; Mean Differences = -278.060, 95% CI 2-sided [-485.2529 to -70.8668], Standard Error of Mean 105.6088
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Daily Activities AUC72; Test type: Superiority or Other; p = 0.013, Piecewise Linear Model; Mean differences = -307.722, 95% CI 2-sided [-551.4006 to -64.0429], Standard Error of Mean 124.1956

34. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) in Work Productivity and Activity (WPAI) Absenteeism Scores Due to Hepatitis C Virus (HCV) Infection and Its Treatment
Description: Time missed from work in hours because of HCV infection or its treatment was assessed by measuring the change from baseline in the Work Productivity and Activity Impairment (WPAI): Hepatitis C questionnaire Absenteeism score (time missed from work, question #2). The number of hours missed from work because of HCV was divided by the total number of hours supposed to work, and expressed as a percentage. An area under the curve (AUC) analysis compared the WPAI absenteeism scores in each treatment group from Baseline to Week 72. The null hypothesis was that there would be no difference between the treatment arms WPAI absenteeism scores from Baseline to Week 72. The Table below shows the lease squares (LS) mean estimates of AUC at Week 72 (as well as at Week 60) in WPAI absenteeism scores and the statistical comparison between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: Analysis Population Description: The intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) was used for all analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 167 | 80
scores on a scale*weeks
  Week 60 | 447.170 [329.8666 to 564.4736] | 400.771 [235.0986 to 566.4429]
  Week 72 | 487.449 [352.1468 to 622.7508] | 430.285 [239.3346 to 621.2359]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Time Missed from Work AUC60; Test type: Superiority or Other; p = 0.642, Piecewise linear model; Mean differences = 46.399, 95% CI 2-sided [-149.6374 to 242.4360], Standard Error of Mean 99.7966
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Time Missed from Work AUC72; Test type: Superiority or Other; p = 0.620, Piecewise Linear Model; Mean differences = 57.164, 95% CI 2-sided [-169.1143 to 283.4414], Standard Error of Mean 115.1548

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Serious Adverse Events (participants affected / at risk) | 10/264 | 8/130
Other Adverse Events (participants affected / at risk) | 252/264 | 124/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=264) | PBO 12Wks PR48 (N=130)
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=264) | PBO 12Wks PR48 (N=130)
Fatigue (General disorders) | 111 | 53
Influenza like illness (General disorders) | 62 | 26
Pyrexia (General disorders) | 51 | 28
Chills (General disorders) | 33 | 18
Asthenia (General disorders) | 25 | 21
Pain (General disorders) | 12 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 68 | 20
Rash (Skin and subcutaneous tissue disorders) | 60 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 33 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 16
Erythema (Skin and subcutaneous tissue disorders) | 15 | 3
Nausea (Gastrointestinal disorders) | 65 | 32
Diarrhoea (Gastrointestinal disorders) | 35 | 19
Vomiting (Gastrointestinal disorders) | 23 | 9
Abdominal pain upper (Gastrointestinal disorders) | 17 | 9
Constipation (Gastrointestinal disorders) | 16 | 4
Dyspepsia (Gastrointestinal disorders) | 14 | 5
Headache (Nervous system disorders) | 88 | 51
Dizziness (Nervous system disorders) | 23 | 9
Dysgeusia (Nervous system disorders) | 16 | 4
Insomnia (Psychiatric disorders) | 56 | 31
Mood altered (Psychiatric disorders) | 39 | 19
Depression (Psychiatric disorders) | 23 | 16
Anxiety (Psychiatric disorders) | 16 | 10
Depressed mood (Psychiatric disorders) | 13 | 11
Sleep disorder (Psychiatric disorders) | 10 | 7
Neutropenia (Blood and lymphatic system disorders) | 54 | 15
Anaemia (Blood and lymphatic system disorders) | 44 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Decreased appetite (Metabolism and nutrition disorders) | 47 | 19
Hyperbilirubinaemia (Hepatobiliary disorders) | 14 | 4
Neutrophil count decreased (Investigations) | 10 | 8
Alanine aminotransferase increased (Investigations) | 3 | 9
Aspartate aminotransferase increased (Investigations) | 3 | 7
Blood thyroid stimulating hormone increased (Investigations) | 1 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days